CLINICAL TRIAL: NCT05563506
Title: The Healthy Kids+ Initiative: Promoting Active Living Through Healthy Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico State University (Other)
Collaborators: Fred Hutch (Unknown)
Responsible Party: Principal Investigator, Dejan Magoc, Assistant Professor, New Mexico State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22769 / 220600102; 2U54CA132383-16 5016 (Other Grant/Funding Number: National Institutes Of Health); 2U54CA132383-16 (NIH)
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Health Behavior
Keywords: physical activity; dietary intake; use of technology; sleep
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Kids + (Experimental): Three times a week for 30 weeks with each session lasting 1 hour.
  Interventions: Behavioral: Healthy Kids +

INTERVENTIONS:
Behavioral: Healthy Kids + — Three times a week for 30 weeks.

SUMMARY:
The study will test the effectiveness and examine the sustained effects of weekly programming on enhancing (1) lifestyle behaviors (physical activity, dietary intake, use of technology, amount of sleep), (2) self-efficacy, (3) self-esteem, and (4) readiness to change among children ages 8-11 years.

DETAILED DESCRIPTION:
The purpose of this study is to implement and evaluate the Healthy Kids+ initiative -- a community-engaged research project - through an existing after-school program in Las Cruces, NM. The Healthy Kids+ initiative will encourage daily lifestyle behaviors (5 or more servings of fruits and vegetables, 2 hours or less of recreational screen time, 1 hour of physical activity, 0 sugary drinks, 10 hours of sleep) that impact childhood obesity. This research project will integrate lessons and activities designed to help kids incorporate changes into their lives to enhance their health and wellness. Overall, it is expected that children participating in the Healthy Kids+ initiative, three times per week, will demonstrate significant changes in improving lifestyle behaviors and maintaining both cognitive and affective changes.Healthy Kids+ will be integrated into the 21st Century afterschool program to provide children at the school sites with relevant PA and health related programming throughout the year. The proposed study will include a repeated-measures research design. A power analysis revealed that for a moderate effect size (f = .25, Cohen, 1988), with five percent type I error and 80% power, three follow up time points, and within subject's correlation of 0.5, we will need to recruit at a minimum 100 total participants. However, our potential participant pool is much larger, and thus we plan on over recruiting (N = 200) to mitigate lost data from attrition rates. The Healthy Kids+ program will be implemented three times a week for 30 weeks. A midyear assessment will be conducted 15-weeks into the program. Participants will then take part in a post assessment at the completion of the 30-week program. The primary quantitative outcome measures include levels of lifestyle behaviors (PA, healthy eating habits, screen time, sleep). The outcome measures will also include self-efficacy, self-esteem, and the level of readiness to change relevant to aforementioned lifestyle behaviors.

Based on Healthy Kids+, we revised and partnered with Fred Hutchinson Cancer Center to expand this trial. For this follow up project, we will recruit 30 children total at NMSU. For this follow up project, we will use accelerometer to objectively measure physical activity and sleep, as well as validated surveys measures for dietary intake and related health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-11 years enrolled in the after-school program at the selected sites.

Exclusion Criteria:

* Children not enrolled in the after-school program at the selected sites.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
After-School Student Questionnaire (ASSQ) | 2 weeks
  A self-administered questionnaire that measures the behavioral and psychosocial variables targeted by the intervention. ASSQ survey items were modified from the Health Behavior Questionnaire and the School-Based Nutrition Monitoring Student Questionnaire, both of which have been found to have acceptable internal consistency (greater than 0.6). Measured constructs in the ASSQ included: food preferences, dietary knowledge, self-efficacy, intentions to choose healthful food options, and participation in sedentary and sports activities.

SECONDARY OUTCOMES:
Children's Sleep Habits Questionnaire (CSHQ) | 1 week
  A parent-rated questionnaire that assesses the frequency of behaviors associated with common pediatric sleep difficulties. A retrospective measure, the CSHQ instructs parents to rate the frequency with which their child has displayed various sleep behaviors during the previous week.
Physical Activity Questionnaire for Children (PAQ-C) | 1 week
  A self-administered, 7-day recall instrument, developed to assess general levels of physical activity for students in grades 4 to 8 and approximately 8 to 14 years of age.

OTHER OUTCOMES:
5-2-1-0 Healthy Habits Questionnaire | 2 weeks
  A brief 10-question survey for children ages 2-14 used to collect information about individuals' healthy habits, specifically habits related to diet, physical activity, screen time, and sleep.
Accelerometer | 2 weeks
  physical activity and sleep
H-PACE Survey | 2 weeks
  demographics, physical activity, dietary intake, screen time, sleep

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Magoc, PhD, Principal Investigator — New Mexico State University; Jason Mendoza, PhD, Principal Investigator — Fred Hutch
Locations (2):
- United States (2):
  - Loma Heights Elementary School, Las Cruces, New Mexico
  - University Hills Elementary, Las Cruces, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data obtained on all standardized measures at baseline and post intervention will be shared with investigators both internal and external to New Mexico State University. Any type of dissemination of results from the project will not identify individual patients. Access levels will be set to protect subject identification and unique identifiers linked to participant identity will be stripped, (i.e., data will be de-identified).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Access will be made available as soon as the primary analyses are completed and accepted for publication in a professional journal and secondary analyses are completed by the team's investigators.
Access Criteria: Prior to sharing the data, Dr. Magoc (PI) will request a detailed plan for data analysis, the choice of the study sample, and a rationale and significance for the proposal. Prior to releasing the data, the proposal will be reviewed by Dr. Magoc.

REFERENCES:
- [Background] Booth M. Assessment of physical activity: an international perspective. Res Q Exerc Sport. 2000 Jun;71(2 Suppl):S114-20. No abstract available. PMID 10925833
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Rovniak LS, Anderson ES, Winett RA, Stephens RS. Social cognitive determinants of physical activity in young adults: a prospective structural equation analysis. Ann Behav Med. 2002 Spring;24(2):149-56. doi: 10.1207/S15324796ABM2402_12. PMID 12054320
- [Background] Steinhardt MA, Dishman RK. Reliability and validity of expected outcomes and barriers for habitual physical activity. J Occup Med. 1989 Jun;31(6):536-46. doi: 10.1097/00043764-198906000-00011. PMID 2786559
- [Background] Kelder S, Hoelscher DM, Barroso CS, Walker JL, Cribb P, Hu S. The CATCH Kids Club: a pilot after-school study for improving elementary students' nutrition and physical activity. Public Health Nutr. 2005 Apr;8(2):133-40. doi: 10.1079/phn2004678. PMID 15877906
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319